CLINICAL TRIAL: NCT02004886
Title: A Multi-Center, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel Panel Study to Assess the Safety, Tolerability and Glucose-Lowering Efficacy of MK-0893 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Assess the Safety, Tolerability and Glucose-Lowering Efficacy of MK-0893 in Participants With Type 2 Diabetes Mellitus (MK-0893-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0893-005
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Therapeutic Uses; Pharmacologic Actions; Molecular Mechanisms of Pharmacological Action; Physiological Effects of Drugs; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — N-((4-(1-(3-(3,5-dichlorophenyl)-5-(6-methoxynaphthalen-2-yl)-1H-pyrazol-1-yl)ethyl)phenyl)carbonyl)-beta-alanine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- MK-0893 (40 mg) (Experimental): MK-0893 40-mg q.d. (quaque die, once daily) group will receive MK-0893 40-mg tablets (after loading dose with 160 mg) and matching placebo to metformin and matching placebo to MK-0893.
  Interventions: Drug: MK-0893; Drug: Placebo
- MK-0893 (120 mg) (Experimental): MK-0893 at 120 mg q.d. group will receive MK-0893 120 mg q.d. tablets (after loading dose of 500 mg on Day 1) and matching placebo tablets to metformin and matching placebo to MK-0893
  Interventions: Drug: MK-0893; Drug: Placebo
- Metformin (2000 mg) (Active Comparator): Metformin taken orally, 500 mg tablets, Day 1 to Day 6: 500 mg b.i.d. (bis in die, twice daily), Day 7 to Day 13: 1000 mg in the morning and 500 mg in the evening, and Day 14 to Day 28: 1000 mg. b.i.d. and matching placebo to MK-0893.
  Interventions: Drug: Metformin; Drug: Placebo
- Placebo (Placebo Comparator): Placebo tablets matching the MK-0893 and placebo tablets matching metformin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-0893 — 10 mg and 100 mg tablets
  Arms: MK-0893 (120 mg); MK-0893 (40 mg)
Drug: Metformin — 500 mg metformin tablets
  Other Names: Glucophage; Glucophage XR; Glumetza; Fortamet; Riomet
  Arms: Metformin (2000 mg)
Drug: Placebo — Placebo tablets matching MK-0893
Drug: Placebo — Placebo tablets matching metformin
  Arms: MK-0893 (120 mg); MK-0893 (40 mg); Placebo

SUMMARY:
This study will assess the safety, tolerability and glucose-lowering efficacy of MK-0893 in participants with type 2 diabetes mellitus. The primary hypothesis is that MK-0893 will reduce 24-hour weighted mean glucose (WMG) significantly more than placebo.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Not currently on antihyperglycemic agent (AHA) or AHA monotherapy (not to include treatment with insulin or thiazolidinediones [i.e., peroxisome proliferator activated receptor-gamma, PPARγ agents])
* male or a female of non-childbearing potential. Women must be postmenopausal or premenopausal and documented surgically sterilized
* A body mass index (BMI) that is > 20 and ≤ 40 kg/m2

Exclusion Criteria:

* History of type 1 diabetes or assessed by the investigator as possibly having type 1 diabetes
* History of ketoacidosis; clinically unstable or rapidly progressive diabetic retinopathy, nephropathy, neuropathy
* Treatment for diabetes within 3 months of study participation with combination anti-hyperglycemic therapy, insulin or thiazolidinediones (e.g., rosiglitazone or pioglitazone)
* oral corticosteroid medications within 2 weeks prior to study participation, or requires digoxin, warfarin, warfarin-like anticoagulants, theophylline, anti-dysrhythmic or anti-seizure medications, immunosuppressants, or anti-neoplastic agents, or herbal remedies
* History of acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV)
* History of gastrointestinal problems or disorders or extensive bowel or gastric surgery
* History of significant or unstable cardiovascular disease
* History of neoplastic disease
* History of hepatic disease
* History of seizures, epilepsy or other neurologic disease
* History of myelodysplastic or pre-leukemic disorders or other severe hematological disorder

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-08-11 (Actual); Primary Completion 2007-02-07 (Actual); Study Completion 2007-02-07 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0893-005&kw=0893-005&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 clinical sites were used in this study in the following countries: Austria, Germany, New Zealand, Russia, and the United States of America.
Groups:
- MK-0893 (40 mg): MK-0893 40-mg, once daily
- MK-0893 (120 mg): MK-0893, 120 mg, once daily
- Metformin (2000 mg): Metformin, oral, 1000 mg, twice daily
- Placebo: Placebo
Period: Overall Study
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Started | 19 | 18 | 18 | 19
Completed | 18 | 17 | 18 | 19
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Unable to attend future visits | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo | Total
Number analyzed (Participants) | 19 | 18 | 18 | 19 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (7.1) | 55.8 (6.8) | 54.7 (8.7) | 51.5 (9.3) | 54.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 12 | 7 | 36
  Male | 11 | 9 | 6 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Weighted Mean Glucose (WMG) at Week 4
Description: Blood samples were collected 30 minutes prior to all meals, and 15, 30, 60, 90, 120, 180 minutes post-meal, then and at midnight, 3 AM, and the next morning at 6:30 AM and 7:30 AM. A 24-hour weighted mean glucose (WMG) was determined by averaging multiple plasma glucose measurements over a 24-hour period.
Time Frame: Baseline and Week 4
Population: Completers Population was used for all efficacy analyses, and required that a participant took at least one dose of study therapy, had a baseline measurement, and had a post-randomization measurement in the treatment period at Week 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 18 | 17 | 18 | 19
mg/dL | -37.9 [-47.1 to -28.8] | -65.7 [-74.8 to -56.5] | -38.1 [-47.0 to -29.2] | -12.0 [-20.7 to -3.4]
Statistical Analysis 1: Comparison: MK-0893 (40 mg) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Terms for treatment, prior AHA therapy status, and baseline 24-hour WMG value as a covariate; Mean Difference (Final Values) = -25.9, 95% CI 2-sided [-38.4 to -13.3]
Statistical Analysis 2: Comparison: MK-0893 (120 mg) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Terms for treatment, prior AHA therapy status, and baseline 24-hour WMG value as a covariate; Median Difference (Final Values) = -53.6, 95% CI 2-sided [-66.1 to -41.1]
Statistical Analysis 3: Comparison: Metformin (2000 mg) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Terms for treatment, prior AHA therapy status, and baseline 24-hour WMG value as a covariate; Mean Difference (Final Values) = -26.0, 95% CI 2-sided [-38.4 to -13.6]

2. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the product.
Time Frame: Up to 42 days
Population: Safety Population included all randomized participants who initiated study therapy.
Measure: Number; unit: Number of Participants
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 19 | 18 | 18 | 19
Number of Participants | 3 | 7 | 9 | 8

3. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the product.
Time Frame: Up to 28 days
Population: Safety Population included all randomized participants who initiated study therapy.
Measure: Number; unit: Number of Participants
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 19 | 18 | 18 | 19
Number of Participants | 0 | 1 | 0 | 0

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Plasma Glucose levels were measured at Baseline and at Week 4. The change from baseline was defined as the Week 4 value minus the Baseline value.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 18 | 17 | 18 | 19
mg/dL | -32.5 [-45.1 to -19.8] | -57.7 [-70.3 to -45.1] | -22.8 [-35.0 to -10.5] | -14.1 [-26.1 to -2.2]
Statistical Analysis 1: Comparison: MK-0893 (40 mg) vs Placebo; Test type: Superiority or Other; p = 0.04, ANCOVA; Relevant baseline efficacy measurements were the covariates; Mean Difference (Final Values) = -18.3, 95% CI 2-sided [-35.7 to -0.9]
Statistical Analysis 2: Comparison: MK-0893 (120 mg) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Relevant baseline efficacy measurements were the covariates; Mean Difference (Final Values) = -43.6, 95% CI 2-sided [-60.9 to -26.3]
Statistical Analysis 3: Comparison: Metformin (2000 mg) vs Placebo; Test type: Superiority or Other; p = 0.320, ANCOVA; Relevant baseline efficacy measurements were the covariates; Mean Difference (Final Values) = -8.6, 95% CI 2-sided [-25.7 to 8.5]

5. Secondary Outcome: Change From Baseline in Fructosamine at Week 4
Description: Fructosamine levels in the blood were measured at Baseline and at Week 4. The change from baseline was defined as the Week 4 value minus the Baseline value.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 18 | 17 | 18 | 19
mg/dL | NA [NA to NA] — Data for this outcome measure were not collected or analyzed. | NA [NA to NA] — Data for this outcome measure were not collected or analyzed. | NA [NA to NA] — Data for this outcome measure were not collected or analyzed. | NA [NA to NA] — Data for this outcome measure were not collected or analyzed.

6. Secondary Outcome: Change From Baseline in Fasting C-peptide at Week 4
Description: Fasting C-peptide levels in the blood were measured at Baseline and at Week 4. The change from baseline was defined as the Week 4 value minus the Baseline value.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 18 | 17 | 18 | 19
ng/mL | 0.1 (0.4) [-0.5 to 0.7] | -0.3 (0.3) [-0.8 to 0.3] | -0.1 (0.3) [-0.6 to 0.5] | -0.0 (0.2) [-0.6 to 0.5]
Statistical Analysis 1: Comparison: MK-0893 (40 mg) vs Placebo; Test type: Superiority or Other; p = 0.751, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.7 to 0.9]
Statistical Analysis 2: Comparison: MK-0893 (120 mg) vs Placebo; Test type: Superiority or Other; p = 0.581, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.0 to 0.6]
Statistical Analysis 3: Comparison: Metformin (2000 mg) vs Placebo; Test type: Superiority or Other; p = 0.918, ANCOVA; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.8 to 0.8]

7. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 4
Description: Fasting insulin levels in the blood were measured at Baseline and at Week 4. The change from baseline was defined as the Week 4 value minus the Baseline value.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: μIU/mL
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 18 | 17 | 18 | 19
μIU/mL | NA [NA to NA] — Data for this outcome measure were not collected or analyzed. | NA [NA to NA] — Data for this outcome measure were not collected or analyzed. | NA [NA to NA] — Data for this outcome measure were not collected or analyzed. | NA [NA to NA] — Data for this outcome measure were not collected or analyzed.

8. Secondary Outcome: Change From Baseline in 2-hour Post-prandial Glucose Excursion at Week 4
Description: 2-hour post-prandial glucose excursion is the change in glucose concentration in the blood 2 hours after a meal. Change from baseline in 2-hour post-prandial glucose excursion at Week 4 is defined as Week 4 minus baseline.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 18 | 17 | 18 | 19
mg/dL | -10.5 [-20.2 to -0.8] | -15.3 [-25.1 to -5.5] | -29.0 [-38.4 to -19.5] | -2.8 [-12.2 to 6.5]
Statistical Analysis 1: Comparison: MK-0893 (40 mg) vs Placebo; Test type: Superiority or Other; p = 0.253, ANCOVA; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-21.1 to 5.6]
Statistical Analysis 2: Comparison: MK-0893 (120 mg) vs Placebo; Test type: Superiority or Other; p = 0.070, ANCOVA; Mean Difference (Final Values) = -12.5, 95% CI 2-sided [-26.0 to 1.0]
Statistical Analysis 3: Comparison: Metformin (2000 mg) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -26.1, 95% CI 2-sided [-39.5 to -12.8]

9. Secondary Outcome: Change From Baseline in 3-hour Area Under the Plasma Concentration Versus Time Curve (AUC) for Glucose at Week 4
Description: Blood samples collected for glucose 30 minutes prior to the breakfast meal and 15, 30, 60, 90, 120, 180 minutes post-meal. AUC is a measure of the amount of drug in the blood over time. 3-hour AUC for Glucose was measured at Baseline and at Week 4. The change from baseline was defined as the Week 4 value minus the Baseline value.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg hr/dL
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 18 | 17 | 18 | 19
mg hr/dL | -128.8 [-169.5 to -88.2] | -230.2 [-270.5 to -189.9] | -136.7 [-175.7 to -97.6] | -39.0 [-77.3 to -0.8]
Statistical Analysis 1: Comparison: MK-0893 (40 mg) vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA; Relevant baseline efficacy measurements were the covariates; Mean Difference (Final Values) = -89.9, 95% CI 2-sided [-145.6 to -34.0]
Statistical Analysis 2: Comparison: MK-0893 (120 mg) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Relevant baseline efficacy measurements were the covariates; Mean Difference (Final Values) = -191.1, 95% CI 2-sided [-246.4 to -135.9]
Statistical Analysis 3: Comparison: Metformin (2000 mg) vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; Relevant baseline efficacy measurements were the covariates; Mean Difference (Final Values) = -97.7, 95% CI 2-sided [-152.4 to -42.9]

10. Secondary Outcome: Change From Baseline in 3-hour AUC for C-peptide at Week 4
Description: Blood samples were collected for C-peptide 30 minutes prior to the breakfast meal and 15, 30, 60, 90, 120, 180 minutes post-meal. AUC is a measure of the amount of drug in the blood over time. 3-hour AUC for C-peptide was measured at Baseline and at Week 4. The change from baseline was defined as the Week 4 value minus the Baseline value.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ng hr/mL
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 18 | 16 | 18 | 18
ng hr/mL | 1.0 [-0.9 to 2.9] | -0.5 [-2.5 to 1.4] | -0.2 [-2.1 to 1.6] | -0.1 [-1.9 to 1.8]
Statistical Analysis 1: Comparison: MK-0893 (40 mg) vs Placebo; Test type: Superiority or Other; p = 0.408, ANCOVA; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-1.5 to 3.7]
Statistical Analysis 2: Comparison: MK-0893 (120 mg) vs Placebo; Test type: Superiority or Other; p = 0.741, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-3.1 to 2.2]
Statistical Analysis 3: Comparison: Metformin (2000 mg) vs Placebo; Test type: Superiority or Other; p = 0.906, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.8 to 2.5]

11. Secondary Outcome: Change From Baseline in 3-hour Insulin Total AUC at Week 4
Description: Blood samples were collected for insulin 30 minutes prior to the breakfast meal and 15, 30, 60, 90, 120, 180 minutes post-meal. AUC is a measure of the amount of drug in the blood over time. 3-hour Insulin Total AUC was measured at Baseline and at Week 4. The change from baseline was defined as the Week 4 value minus the Baseline value.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: µIU hr/mL
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Number analyzed (Participants) | 17 | 15 | 18 | 19
µIU hr/mL | 5.3 [-15.5 to 26.1] | 6.1 [-15.3 to 27.6] | 1.2 [-18.4 to 20.7] | 7.8 [-11.2 to 26.8]
Statistical Analysis 1: Comparison: MK-0893 (40 mg) vs Placebo; Test type: Superiority or Other; p = 0.857, ANCOVA; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-30.4 to 25.3]
Statistical Analysis 2: Comparison: MK-0893 (120 mg) vs Placebo; Test type: Superiority or Other; p = 0.906, ANCOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-30.3 to 26.9]
Statistical Analysis 3: Comparison: Metformin (2000 mg) vs Placebo; Test type: Superiority or Other; p = 0.630, ANCOVA; Mean Difference (Final Values) = -6.6, 95% CI 2-sided [-34.0 to 20.8]

ADVERSE EVENTS:
Time Frame: Up to 42 days
Description: Safety Population included all randomized participants who initiated study therapy. Adverse events were collected up to 14 days after last dose of study drug.
Arm/Group | MK-0893 (40 mg) | MK-0893 (120 mg) | Metformin (2000 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 3/19 | 7/18 | 9/18 | 8/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-0893 (40 mg) (N=19) | MK-0893 (120 mg) (N=18) | Metformin (2000 mg) (N=18) | Placebo (N=19)
External Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 1 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 3 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Gingival Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Stomach Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1
Feeling Abnormal (General disorders) | 0 | 1 | 0 | 0
Nodule (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1
Herpes Simplex (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 2
Otitis Media (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 1 | 1 | 0 | 1
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Testicular Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.